CLINICAL TRIAL: NCT05548335
Title: Microconvex Probe Versus Linear Probe for Measurement of the Optic Nerve Sheath Diameter
Brief Title: Measurement of the Optic Nerve Sheath Diameter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cleveland Clinic Akron General (Other)
Responsible Party: Principal Investigator, Joshua Jacquet, Physician, Cleveland Clinic Akron General
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21036
Record Dates: First submitted 2022-07-01; First posted 2022-09-21 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Optic Nerve
Keywords: ocular ultrasound; optic nerve sheath diameter; ETD

STUDY DESIGN:
Intervention Model Description: There are no groups. All subjects will have the same inclusion criteria and will have the same intervention.
Masking Description: No masking. All subjects have same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocular Ultrasound (Other): This arm includes all patients enrolled who will have an ocular ultrasound with two different probes for a total of four ultrasounds.
  Interventions: Procedure: Ocular Ultrasound

INTERVENTIONS:
Procedure: Ocular Ultrasound — 1. Patients presenting to the emergency department and have a normal head and/or ocular computed tomography scan will be considered for inclusion in this study. Study staff will discuss the study with the patient and obtain consent. At that point, operator will perform ocular ultrasound. Procedure will start with either the linear or microconvex probe. A single-use sterile gel packet will be used to apply gel to one closed eyelid. The probe will be placed with minimal pressure on the eye. A transverse measurement of the ONSD will be taken. In this same view the maximal transverse diameter of the eyeball will also be measured. Images of the eye with ONSD and ETD measurements will be captured. Repeat until three measurements have been obtained resulting in an average ONSD and ETD for that eye. Repeat for other eye. Switch probe and repeat on both eyes.

SUMMARY:
This study is a prospective assessment of the accuracy of ocular ultrasound as a tool to measure the diameter of the optic nerve sheath and the eyeball transverse diameter in healthy adult patients presenting to the Emergency Department and have confirmatory imaging of the optic nerve as part of their clinical care.

DETAILED DESCRIPTION:
This will be a prospective evaluation of accuracy of microconvex and linear transducers for ultrasound measurements of the ONSD and the ETD. Study population will be adult patients that present to Cleveland Clinic Akron General Emergency Department between July 1, 2022 and July 31 April 1, 2023. Patients will be identified on the Emergency Medicine Department tracking board. Patients, once identified as meeting inclusion criteria will be asked to participate in this study and full written consent will be required. All participants will have identical procedures and there will be no groups.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age and older, and;
* Present to Cleveland Clinic Akron General's ED (Main)
* Have CT head and/or ocular ordered as a part of clinical care that is read as normal or no acute disease (confirmatory imaging), and;
* Agree to and provide written consent for participation.

Exclusion criteria:

* Acute ocular pathology
* Abnormal brain and/or ocular CT
* History of increased intracranial pressure or optic nerve disease
* Not medically stable
* Pregnant or incarcerated
* Unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Primary objective is to determine the accuracy of the microconvex ultrasound transducer as compared to the linear ultrasound transducer for ultrasound measurement of the optic nerve sheath diameter compared to CT measurements. | through study duration, one year is anticipated.
  The patient will be enrolled and be involved with the study for 15-20 minutes. At this time the research procedures will be done.

SECONDARY OUTCOMES:
To determine the level of intra- and inter-rater variability for ultrasound measurement of the optic nerve sheath diameter between the two transducer types. | through study duration, one year is anticipated.
  The patient will be enrolled and be involved with the study for 15-20 minutes. At this time the research procedures will be done.
To determine the accuracy of the microconvex ultrasound transducer as compared to the linear ultrasound transducer for ultrasound measurement of the eyeball transverse diameter compared to CT measurements. | through study duration, one year is anticipated.
  The patient will be enrolled and be involved with the study for 15-20 minutes. At this time the research procedures will be done.
To determine the accuracy of the microconvex ultrasound transducer as compared to the linear ultrasound transducer for ultrasound measurement of the ONSD/ETD compared to CT measurements. | through study duration, one year is anticipated.
  The patient will be enrolled and be involved with the study for 15-20 minutes. At this time the research procedures will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Jacquet, MD, Principal Investigator — Cleveland Clinic Akron General
Locations (1):
- Cleveland Clinic Akron General, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No